CLINICAL TRIAL: NCT02474667
Title: A Multicenter, Prospective, Double-Blind, Randomized, Placebo-Controlled, Phase 3 Study of ANG-3777 (Formerly BB3) to Improve Graft Function and Reduce the Severity of Kidney Dysfunction or Delayed Graft Function Following Kidney Transplantation in Recipients of a Deceased Donor Kidney
Brief Title: Reduce the Severity of DGF in Recipients of a Deceased Donor Kidney
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Angion Biomedica Corp (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001-15
Record Dates: First submitted 2015-06-12; First posted 2015-06-18 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-04

CONDITIONS: Delayed Graft Function
Keywords: DGF; Delayed Graft Function; Renal Transplantation; Deceased Donor Kidney; BB3; Kidney Transplantation; Acute Kidney Injury
MeSH Terms: conditions — Delayed Graft Function; Acute Kidney Injury | interventions — terevalefim; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BB3 (Active Comparator): Administered IV for 30 min within 24 hours after transplantation and around 24 hours after previous dosing 3 days in a row
  Interventions: Drug: ANG-3777
- Normal Saline (Placebo Comparator): Administered IV for 30 min within 24 hours after transplantation and around 24 hours after previous dosing 3 days in a row
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ANG-3777
  Other Names: Hepatocyte growth factor mimetic; BB3
  Arms: BB3
Other: Placebo
  Other Names: Normal saline
  Arms: Normal Saline

SUMMARY:
The major objective is to demonstrate the safety and efficacy of ANG-3777 in improving graft function and reducing the severity of delayed graft function (DGF) in recipients at high risk of DGF after receiving a deceased donor renal allograft.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must provide written informed consent using an Institutional Review Board/Independent Ethics Committee (IRB/IEC) approved consent form, and must understand and be willing and able to comply with the requirements of the study, including screening procedures and all required study visits.
2. Males and females ≥ 18 years of age.
3. Renal failure requiring hemodialysis or peritoneal dialysis initiated at least 3 months prior to transplantation.
4. Patient is to be the recipient of a first kidney transplant from a deceased donor.
5. Study drug can be administered starting within 30 hours after restoration of blood flow to the engrafted kidney.
6. Body mass index < 40 based on dry weight. Dry weight and height parameters obtained within 7 days prior to study entry may be used..
7. Estimated donor organ cold ischemia time less than 30 hours (for PMP kidneys less than 40 hours).

Exclusion Criteria

1. Scheduled for multiple organ transplantation or prior recipient of a transplanted organ.
2. Recipient of an ABO-incompatible kidney.
3. Recipient of pediatric en-bloc kidney transplantation or adult or pediatric planned transplant of dual kidneys (from the same donor) not transplanted en bloc.
4. Recipient of a kidney preserved by normothermic pulsatile machine perfusion.
5. Has measurable donor-specific antibody or positive cross-match requiring desensitization prior to transplantation or deviation from standard immunosuppressive therapy.
6. Currently participating in or has participated in an investigational drug or medical device study within 30 days or five drug half-lives, whichever is longer, prior to enrollment into this study. Patients cannot be given another investigational agent during the course of this study (through Day 360). Patients may participate in another concurrent study only if that study is a non-interventional, observational investigation.
7. Concurrent sepsis or active bacterial infection.
8. Has an active malignancy or history within 5 years prior to enrollment in the study, of solid, metastatic or hematologic malignancy with the exception of basal or squamous cell carcinoma in situ of the skin that has been adequately treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
The severity of DGF | Day 360
  The primary endpoint is renal function assessed by eGFR (using the CKD-EPI equation based on serum creatinine), with a primary analysis time point consisting of eGFR at month 12.

CONTACTS AND LOCATIONS:
Overall Officials: John Neylan, MD, Study Director — Angion Biomedica
Locations (30):
- United States (30):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Keck Hospital of USC, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - California Institute of Renal Research, San Diego, California
  - California Pacific Medical Center (Sutter), San Francisco, California
  - University of California San Francisco Medical Center, San Francisco, California
  - University of Colorado Hospital Anschuts Medical Campus, Aurora, Colorado
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Rush University, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - Kansas University, Lawrence, Kansas
  - University of Louisville, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center BRANY, The Bronx, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Houston Methodist Hospital, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University (VCU) Medical Center of Virginia, Richmond, Virginia
  - University of Washinton Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin